CLINICAL TRIAL: NCT06001138
Title: FutureMS-2: Clinical, Laboratory, and Genomic Predictors of Disease Activity in People Diagnosed With Relapsing Onset Multiple Sclerosis: an Observational Cohort and Scottish Precision Medicine Study
Brief Title: Multiple Sclerosis: FutureMS-2 - an Observational Cohort and Scottish Precision Medicine Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC21029
Record Dates: First submitted 2023-02-07; First posted 2023-08-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FutureMS is a project created in direct response to frequent questions people with MS ask their doctors. Every person newly diagnosed wants to know how MS will affect them over their life and what can be done to stop the disease progressing and improve their quality of life. FutureMS aims to help answer those questions.

The original FutureMS study provided a snapshot of the impact of MS within a year of diagnosis. However, MS is a long-term condition and so the investigators now want to better understand the impact of MS, on the same individuals, after approximately 5 and 10 years of living with MS. This is the purpose of FutureMS-2.

DETAILED DESCRIPTION:
MS is a chronic incurable and devastating inflammatory - neurodegenerative disorder of the central nervous system. There are an estimated 2.4M people with multiple sclerosis (pwMS). Scotland has one of the highest prevalence for MS in the world with 240 per 100'000 of the population having MS at any given time and with an incidence rate of 8.76 per 100'000. It is the leading non-traumatic cause of neurological disability in young adults across the industrialised world, and 85% of prevalent cases are in people of working age.

Despite important advances in diagnostics and treatment for the newly diagnosed pwMS, there remain major unsolved challenges. These include the inability to predict disease course and prognosis for newly diagnosed patients. MS in this regard is distinct to other degenerative brain diseases that have a uniform and predictable "downward" natural history. In contrast, MS is inherently unpredictable and variable. For example, some pwMS will, without treatment, experience a mild course with negligible disability after many years whilst others are seriously disabled within a few years. Therefore, at the point of diagnosis of MS, today the investigators are unable to predict whether the individual is destined to have mild, intermediate or a severe disease course noting that the disease is chronic and plays out over 30+ years. Furthermore, the range of disabilities that pwMS endure are varied and many and extend beyond physical disability. Yet, "invisible" but devastating disability including fatigue, pain and cognition, remain poorly studied and understood. As a consequence of these knowledge gaps, pwMS are unable to make informed lifestyle or treatment decision choices. FutureMS aims to address these important knowledge gaps.

Against this background, FutureMS supported by SMS Scotland was established (2015 - 2021). FutureMS is a national inception cohort study of 440 newly diagnosed people with MS that combines clinical, imaging, genomic, health and lifestyle data using a Scottish informatics platform. FutureMS is very much a key plank of the wider ambition for Scotland to lead in the area of precision medicine with a special focus on disorders, such as MS, with high morbidity and cost to the individual and society. Scotland is ideally placed to lead in precision medicine for MS. This reflects disproportionate per capita disease burden plus various national assets including e-health infrastructural strengths, unitary single health provider, single health identifier and 5 research intensive medical universities with many world-leading researchers in both the laboratory and clinical science of MS. Many of these researchers are also investigators in the MS Society Centre of Excellence - one of only two UK flagship centres supported by the MS Society - based in Edinburgh (Director - Siddharthan Chandran).

Next phase for FutureMS - Wave 2. The ultimate objective of FutureMS-2 is to contribute to the generation of validated and quantitative precision medicine tools that will allow individualised disease course prediction and personalised treatment. To fully exploit this national resource and realise its unprecedented value, there is a need to follow up the FutureMS cohort over time and "re-measure" key metrics of disease activity and its impact on the health and wealth of the individual. The wider goals of Wave 2 are to further drive the agenda and ambition of 4Ps (prevent, personalise, predict and participate) medicine for MS. It is the investigators' intention to grow, in particular, the "participatory" elements of this programme working with and advised/guided by the FutureMS "lived experience panel". This study has been shaped by these discussions and details the scientific justification and methodology to allow two follow up epochs of the original cohort at c.5 years (Wave 2) and c.10 years after diagnosis (Wave 3). Eight-ten years is the approximate average time by which the majority of individuals, without treatment, with RRMS will transition to the progressive phase of MS.

ELIGIBILITY:
Inclusion Criteria:

* Previous participants in FutureMS cohort
* Capacity to provide informed consent

Exclusion Criteria:

* Not a participant of FutureMS inception cohort
* Contraindication to MR brain imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The overwhelming majority (98%) of FutureMS participants have given consent to be approached for future research. The study aims to retain 90% of the consented FutureMS cohort. The majority of participants that took part in FutureMS gave their consent to be contacted about future ethically approved research. These participants will be contact directly by a phone, email or post by the study team.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Disease activity defined by new or enlarging T2 hyperintense lesion count on MR brain imaging at 5 years and 10 years of diagnosis with relapsing-remitting MS | at 5 and 10 years after diagnosis of relapsing - remitting MS
  Primary objective

SECONDARY OUTCOMES:
Disease activity defined by the composite endpoint of new or enlarging T2 hyperintense lesions on MR brain imagingneurodegeneration and regenerative markers of disease activity | at 5 and 10 years after diagnosis of relapsing - remitting MS
  Co-secondary outcome
clinical relapse at 5 and 10 years of diagnosis with relapsing-remitting MS | at 5 and 10 years after diagnosis of relapsing - remitting MS
  Co-secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Siddharthan Chandran, Professor, Study Director — University of Edinburgh
Locations (5):
- United Kingdom (5):
  - Aberdeen Clinical Research Facility Royal Cornhill Hospital, Aberdeen
  - Dundee Clinical Research Centre Ninewells Hospital, Dundee
  - Anne Rowling Regenerative Neurology Clinic, Edinburgh
  - Glasgow Clinical Research Facility Queen Elizabeth University Hospital, Glasgow
  - Centre for Health Sciences Raigmore Hospital, Inverness

IPD SHARING:
Plan to Share IPD: Yes
To ensure data transparency, the results of any closed comparisons will be published in a peer reviewed journal as soon as it is possible when the integrity of the study will not be affected.
  Individual level participant data will be shared, after de-identification, upon receipt of a valid request.
  Some data may be shared prior to the publication of study results depending on the requirements, however, no end point data will be released without explicit need.
  Each data request form will be individually reviewed to ensure the proposal has a valid rationale and appropriate methodology. Only data required for the project will be shared.
  A summary of results will be provided to all participants via newsletters and the Anne Rowling Clinic's website.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of study results, no end date.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims of the proposal only.
  Data sharing request forms are available from future-ms@ed.ac.uk. Requesters will need to sign a data access agreement prior to being provided with access to data.

REFERENCES:
- [Background] Kearns PKA, Martin SJ, Chang J, Meijboom R, York EN, Chen Y, Weaver C, Stenson A, Hafezi K, Thomson S, Freyer E, Murphy L, Harroud A, Foley P, Hunt D, McLeod M, O'Riordan J, Carod-Artal FJ, MacDougall NJJ, Baranzini SE, Waldman AD, Connick P, Chandran S. FutureMS cohort profile: a Scottish multicentre inception cohort study of relapsing-remitting multiple sclerosis. BMJ Open. 2022 Jun 29;12(6):e058506. doi: 10.1136/bmjopen-2021-058506. PMID 35768080